CLINICAL TRIAL: NCT03308981
Title: Efficacy of the REThink Therapeutic Online Game in Promoting Child and Adolescent Mental Health
Brief Title: Efficacy of the REThink Therapeutic Online Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: Romanian National Authority for Scientific Research (Unknown)
Responsible Party: Principal Investigator, Oana David, Associate Professor Oana David, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REThink therapeutic game
Record Dates: First submitted 2017-09-27; First posted 2017-10-13 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Resilience, Psychological
Keywords: therapeutic online game; resilience; prevention; emotional disorders; child; adolescent

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three groups: 1) REThink group, 2) Rational-Emotive-Behavioral Education (REBE) group and 3) wait-list condition.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- REThink therapeutic online game (Experimental): REThink group will play twice the seven levels of the game, divided into seven modules.
  Interventions: Device: REThink therapeutic online game
- REBE group (Active Comparator): Participants will follow 7 modules, structured based on the strategies practiced in each of the REThink level.
  Interventions: Other: REBE group
- Wait-list (No Intervention): Participants will not receive any intervention.

INTERVENTIONS:
Device: REThink therapeutic online game — The REThink therapeutic online game has seven levels. Each level has various degrees of complexity, which increase as the player progresses in the game. The scenario of the game was developed based on the REBT model, such that it focuses on: a. identifying the emotional and behavioral reactions; b. identifying cognitive processes; c. identifying the relation between cognitive processes and emotions and behavioral reactions; d. changing irrational cognitions into rational cognitions; e. building problem solving skills; f. building relaxation skills and g. building happiness skills.
  Arms: REThink therapeutic online game
Other: REBE group — In the Rational-Emotive-Behavioral Education (REBE) group participants will follow 7 modules, structured based on the strategies practiced in each of the REThink level.
  Arms: REBE group

SUMMARY:
This study aims to test the efficacy of the REThink therapeutic online video game. Children and adolescents (N = 150), aged between 10-16 years, will be randomly assigned to one of three groups: 1) REThink group, 2) Rational-Emotive-Behavioral Education (REBE) group and 3) wait-list condition.

DETAILED DESCRIPTION:
Background:The prevalence of emotional disorders in children and adolescents is constantly growing and leads to long-term negative consequences for later functioning. An efficient way to approach emotional disorders in youths is to provide adequate services to them prior to the onset of symptoms. A new strategy for implementing prevention programs in youths is the use of therapeutic games. The aim of this study is to test the effectiveness of the REThink therapeutic online game,in helping children and adolescents, aged between 10-16 years, to develop psychological resilience.

Methods: To test the effectiveness of the REThink therapeutic online game, 150 children and adolescents aged between 10-16 years will be included in the study. Participants will be randomly assigned to one of three groups: 1) the online therapeutic game intervention (REThink group), 2) the control condition Rational-Emotive-Behavioral Education (REBE) group and 3) the wait-list condition. Participants in the REThink group will play the seven levels of the game, structured into seven modules. In the REBE group, participants will follow seven REBE lessons, structured based on the strategies practiced in each of the REThink level. Assessment of participants will be made before, at the middle, at the end of the intervention, and at 6 months after the intervention.

Results: It is expected that participants in the REThink group will provide significantly better results regarding primary outcomes, namely psychological adjustment and the intensity of emotions. Significant improvements are expected at post-test and follow up for the REThink group regarding secondary outcomes, emotion regulation skills, temperamental variables, anxiety in a stressful situation, problem solving skills, relaxation skills,and alpha asymmetry index, compared to wait-list condition, and similarly to the REBE group. Also, it is expected that REThink efficacy will be related to changes in irrational beliefs, and negative and positive automatic thoughts. In addition, it is expected that the REThink game will register high satisfaction with the intervention.

Conclusions: This is randomized controlled trial which aims to analyze the effectiveness of a new therapeutic game developed for children and adolescents will provide important information regarding this promising tool.

ELIGIBILITY:
Inclusion Criteria:

* aged between 10-16 years
* provided written parental consent

Exclusion Criteria:

* Intellectual disability or physical limitations precluded the use of the computer program
* Had a major mental health disorder
* Had had (in past three months) or was having psychotherapy or psychiatric treatment

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Emotional symptoms | 12 months
  Strengths and Difficulties Questionnaire - child version (SDQ; Goodman, 1997)
Depressed mood | 12 months
  The Early Adolescent Temperament Questionnaire - Revised (EATQ-R; Ellis, 2002)

SECONDARY OUTCOMES:
Emotion-regulation | 12 months
  The Emotion Regulation Index for Children and Adolescents (ERICA; Biesecker & Easterbrooks, 2001)
Temperament | 12 months
  The Early Adolescent Temperament Questionnaire - Revised (EATQ-R; Ellis, 2002) contains 65 questions in the self-report form and is designed to measure temperamental effortful control, affiliativeness, surgency, and negative affectivity. We will use in the present study only 4 subscales from the original questionnaire: attention, fear, inhibitory control and depressive mood.
Negative and positive emotions | 12 months
  The Functional and Dysfunctional Child Mood Scales (David & DiGiuseppe, 2016) is used in the game having included faces of children that appear during the game levels. The scale is new and will be used cautiously since only preliminary data is available concerning its psychometrics.
Satisfaction with the intervention | 12 months
  Treatment Satisfaction Visual Analogue Scales-TS-VAS (Zecca et al., 2014)

OTHER OUTCOMES:
Irrational beliefs | 12 months
  The Child and Adolescent Scale of Irrationality (CASI; Bernard & Cronan, 1999) will be used to measure irrational cognitions in children and adolescents, a hypothesized mediating variable.
Automatic Thoughts | 12 months
  Children's Automatic Thoughts Scale-Negative/Positive (CATS-N/P; Hogendoorn et al., 2010) is a 50-item questionnaire that assesses negative and positive automatic thoughts in children and adolescents. This variable is a hypothesized mediating variable.
Anxiety in a stressful situation | 12 months
  The Profile of Affective Distress (PDA; Opriș & Macavei, 2007)
Frontal alpha asymmetry | 12 months
  EMOTIV Epoc+ (www.emotiv.com) will measure frontal brain activity at rest and during a stressful task at pre-post and follow-up.
Heart rate | 12 months
  Polar Heart Rate Sensor (http://www.polar.com) will measure heart rate in a stressful situation pre, post and at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Oana A David, PhD, Study Director — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Faculty of Psychology and Educational Sciences, Department of Clinical Psychology and Psychotherapy, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] David OA, Fodor LA. Are gains in emotional symptoms and emotion-regulation competencies after the REThink therapeutic game maintained in the long run? A 6-month follow-up. Eur Child Adolesc Psychiatry. 2023 Oct;32(10):1853-1862. doi: 10.1007/s00787-022-02002-w. Epub 2022 May 20. PMID 35593966
- [Derived] David OA, Cardos RAI, Matu S. Is REThink therapeutic game effective in preventing emotional disorders in children and adolescents? Outcomes of a randomized clinical trial. Eur Child Adolesc Psychiatry. 2019 Jan;28(1):111-122. doi: 10.1007/s00787-018-1192-2. Epub 2018 Jul 10. PMID 29992353
- [Derived] David OA, Cardos RAI, Matu S. Changes in irrational beliefs are responsible for the efficacy of the REThink therapeutic game in preventing emotional disorders in children and adolescents: mechanisms of change analysis of a randomized clinical trial. Eur Child Adolesc Psychiatry. 2019 Mar;28(3):307-318. doi: 10.1007/s00787-018-1195-z. Epub 2018 Jul 9. PMID 29987559